CLINICAL TRIAL: NCT04749849
Title: Sedentary Behavior, Physical Activity, Sleep, and Cardiovascular Risk in Pregnancy: the Pregnancy 24/7 Cohort Study
Brief Title: The Pregnancy 24/7 Cohort Study
Status: Completed | Type: Observational
Sponsor: Kara Whitaker (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pittsburgh (Other); West Virginia University (Other)
Responsible Party: Sponsor-Investigator, Kara Whitaker, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202002630; R01HL153095 (NIH)
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications; Sedentary Behavior; Physical Activity; Sleep
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Moderate to vigorous intensity physical activity is known to reduce the risk of hypertensive disorders of pregnancy and other adverse pregnancy outcomes that increase future maternal cardiovascular disease risk (2018 Physical Activity Guidelines Advisory Committee, 2018; Davenport et al., 2018), yet less than 25% of pregnant women meet public health physical activity guidelines (Hesketh & Evenson, 2016). More than 95% of the 24-hour day is spent in sedentary behavior, sleep, or light-intensity activity; however, the impacts of these lower intensity activities on adverse pregnancy outcomes are unknown. This multi-site observational cohort study (N=500) will leverage state-of-the-art, 24-hour behavior assessment in each trimester of pregnancy and examine associations with adverse pregnancy outcomes to inform guidelines and future interventions designed to improve women's pregnancy and long-term cardiovascular health.

DETAILED DESCRIPTION:
The overall goal of this study is to use state-of-the-art monitors to objectively measure the 24-hour behavioral cycle (sedentary behavior, sleep, and physical activity) in each trimester of pregnancy, and to examine associations of these behaviors with hypertensive disorders of pregnancy and other adverse pregnancy outcomes linked with future cardiovascular disease (CVD) risk. For this, 500 women in early pregnancy will be recruited to take part in a multi-site (Universities of Iowa and Pittsburgh) cohort study. Women will wear two state-of-the-art devices for seven days in each trimester of pregnancy to assess sedentary behavior and physical activity (activPAL micro 3) as well as sleep (ActiWatch Spectrum Plus). Hypertensive disorders of pregnancy and other adverse outcomes will be obtained through medical chart abstraction. This project will inform guidelines on optimal 24-hour behavioral patterns in pregnancy, as well as lay the foundation for future studies testing behavioral interventions in pregnancy to achieve optimal outcomes and improve women's long-term cardiovascular health.

Specific Aims:

AIM 1: Examine associations of sedentary behavior patterns with hypertensive disorders of pregnancy. Hypothesis: Women with a consistently high sedentary behavior pattern across trimesters will have higher incidence of gestational hypertension/preeclampsia, after adjustment for MVPA.

AIM 2: Examine associations of sleep patterns with hypertensive disorders of pregnancy. Hypothesis: Women with short sleep duration or poor sleep quality patterns across trimesters will have higher incidence of gestational hypertension/preeclampsia, after adjustment for MVPA.

AIM 3: Determine optimal 24-hour behavioral patterns during pregnancy to reduce the risk of hypertensive disorders of pregnancy. Hypothesis: Statistically reallocating time in sedentary behavior for LPA or MVPA, but not sleep (among adequate duration sleepers), will be associated with lower incidence of gestational hypertension/preeclampsia.

Significance: Pregnancy is a critical period for future cardiovascular health where unmasked cardiovascular disease (CVD) risk factors contribute to the development of maternal CVD later in life (Catov, 2015). The American Heart Association (AHA) now recognizes adverse pregnancy outcomes, including gestational hypertension and preeclampsia as key risk factors for CVD (Mosca et al., 2011). CVD remains the leading cause of mortality among women in the United States, accounting for one-third of all deaths (Benjamin et al., 2018). Stagnant CVD rates in young women are a particular public health problem. While overall CVD mortality rates have decreased over the last 20 years, mortality rates in women younger than 55 years have plateaued (Benjamin et al., 2018; Wilmot, O'Flaherty, Capewell, Ford, & Vaccarino, 2015). In order to reduce the burden of CVD, it is essential to focus on populations who are more likely to develop CVD risk factors, including women of reproductive age. Identifying modifiable behavioral factors that are associated with adverse pregnancy outcomes could help prevent these conditions and the long-term risk they bring to women.

Based on guidelines, women during pregnancy should generally 'move more and sit less' throughout the day (2018 Physical Activity Guidelines Advisory Committee, 2018). While there is currently insufficient evidence to define specific quantitative targets for limiting sedentary behavior in the general population or pregnant women, the 2018 Physical Activity Guidelines Advisory Committee highlighted sedentary behavior and pregnancy as two key topics in need of further research. The American College of Obstetricians and Gynecologists (ACOG) also does not have sedentary behavior guidelines during pregnancy, although growing evidence suggests prescribed bed rest may actually increase the risk of adverse pregnancy outcomes, rather than decreasing risk as previously thought (Matenchuk et al., 2019). Guidelines also suggest that pregnant women should sleep 7 to 9 hours per night on a regular basis (Watson et al., 2015). Yet, uncertainty remains about the health effects of short or long sleep duration during pregnancy, as well as how sleep quality influences pregnancy outcomes.

In Aim 1, the proposed research will inform quantitative guidelines for sedentary behavior patterns and the development of cardiovascular risk during pregnancy. Aim 2 will address existing gaps by evaluating objectively-measured sleep quantity and quality to understand nuances in sleep across pregnancy and implications for health outcomes. As established guidelines recommend pregnant women get 150 minutes of aerobic MVPA per week or approximately 20-30 minutes per day, this is not the focus of the current study. However, MVPA is an important component of the 24-hour behavioral cycle and must be assessed to understand which 24-hour behavioral patterns are most associated with optimal cardiovascular health during pregnancy, as proposed in Aim 3. Our primary outcome of interest is hypertensive disorders that develop during pregnancy (gestational hypertension and preeclampsia) given the high and rising prevalence of these conditions, strong association with future maternal CVD, and promising pilot data indicating that sedentary behavior may be associated with these conditions, even after adjustment for MVPA.

Examining the dynamic interplay of sedentary behavior, sleep, and physical activity (conceptualized as a 24-hour behavioral cycle) is critical to determine optimal patterns for pregnancy health. Given that there is a finite amount of time in a day, increasing time in one behavior requires decreasing time in another behavior. The effects of sedentary behavior, sleep, and physical activity on health outcomes are not only dependent on each behavior, but also on the behavior that they displace (Mekary, Willett, Hu, & Ding, 2009). While these behaviors are often studied in isolation, this new paradigm considers the importance of examining the combined role of sedentary behavior, sleep, and physical activity on health outcomes (Buman et al., 2014). Emerging statistical methods to test hypotheses within finite time constraints will allow us to better understand the full 24-hour behavioral cycle and how these activity domains can be coupled and leveraged for health promotion and disease prevention. This study will address a critical gap in knowledge by examining how the 24-hour behavioral cycle is related to hypertensive disorders of pregnancy or other adverse outcomes that increase CVD risk.

In summary, preventing hypertensive disorders of pregnancy and other adverse outcomes is a potentially potent public health approach to reduce the burden of CVD in women. In the context of increasing incidence and limited treatment options, there is a critical need to identify novel, modifiable intervention targets that could prevent adverse pregnancy outcomes and improve women's cardiovascular health.

ELIGIBILITY:
Inclusion:

Adult subjects inclusion criteria:

* Pregnant, <13 weeks gestation
* 18-45 years of age

Exclusion:

Adult subjects exclusion criteria:

* Taking medications for hypertension or diabetes
* Medical condition that severely limits physical activity (cannot walk ½ mile or climb 2 flights of stairs)
* Undergoing treatment for sleep disorders (medication, behavioral treatment, or mechanical therapies)
* Other serious medical condition (such as systemic lupus, chronic renal disease, hepatitis)

Minor subjects inclusion criteria:

• Mother took part in the Pregnancy 24/7 Study and consented to medical chart abstraction of child

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in their first trimester of pregnancy (10 weeks 0 days - 12 weeks 6 days gestation) who complete eligibility screening: 250 from the Iowa site, 125 from the Pittsburgh site, and 125 from the West Virginia site
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Hypertensive disorders of pregnancy | Through study completion for each participant, an average of 7.5 months after enrollment
  Gestational hypertension and preeclampsia, assessed through medical chart review

SECONDARY OUTCOMES:
Gestational diabetes | Through study completion for each participant, an average of 7.5 months after enrollment
  Assessed through medical chart review
Preterm delivery | At study completion for each participant (delivery), an average of 7.5 months after enrollment
  Defined as delivery <37 weeks gestation, assessed through medical chart review
Low birth weight | At study completion for each participant (delivery), an average of 7.5 months after enrollment
  Defined as birthweight<10th percentile for gestational age, assessed through medical chart review
All adverse pregnancy outcomes (composite) | Through study completion for each participant, an average of 7.5 months after enrollment
  Composite measure including gestational hypertension, preeclampsia, gestational diabetes, preterm delivery, and low birth weight, assessed through medical chart review
Blood pressure | Through study completion for each participant, an average of 7.5 months after enrollment
  Assessed during the first trimester study visit and through medical chart review
Glycemic control | Through study completion for each participant, an average of 7.5 months after enrollment
  From glucose tolerance test, assessed through medical chart review

CONTACTS AND LOCATIONS:
Overall Officials: Kara Whitaker, PhD, MPH, Principal Investigator — University of Iowa; Bethany Barone Gibbs, PhD, Principal Investigator — West Virginia University; Christopher Kline, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Bethany Barone Gibbs, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified data that are relevant to the primary aims of the study will be made available along with a relevant data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible, no later than the time of an associated publication, or the end of the award period, whichever comes first.
Access Criteria: Data access will be provided to external researchers who provide a methodologically sound proposal for secondary data analysis that is approved by the investigators of the study. Proposals should be directed to the study PI.

REFERENCES:
- [Background] Nuckols VR, Davis KG, Pierce GL, Gibbs BB, Whitaker KM. Associations of physical activity and sedentary time with aortic stiffness and autonomic function in early pregnancy. J Appl Physiol (1985). 2025 Mar 1;138(3):774-782. doi: 10.1152/japplphysiol.00889.2024. Epub 2025 Feb 14. PMID 39951544
- [Background] Kozai AC, Jones MA, Borrowman JD, Hauspurg A, Catov JM, Kline CE, Whitaker KM, Gibbs BB. Patterns of physical activity, sedentary behavior, and sleep across pregnancy before and during two COVID pandemic years. Midwifery. 2025 Feb;141:104268. doi: 10.1016/j.midw.2024.104268. Epub 2024 Dec 18. PMID 39721225
- [Background] Gallagher JB, Boonstra DE, Borrowman JD, Unke M, Jones MA, Kline CE, Barone Gibbs B, Whitaker KM. Comparing Multiple Approaches to Estimate Physical Activity, Sedentary Behavior, and Sleep in Pregnancy. J Meas Phys Behav. 2024 Jan;7(1):jmpb.2024-0007. doi: 10.1123/jmpb.2024-0007. Epub 2024 Nov 19. PMID 39949639
- [Background] Gibbs BB, Jones MA, Whitaker KM, Ross ST, Davis KK. Measurement of Barriers, Attitudes, and Expectations for Sitting Less in Pregnancy. Am J Health Behav. 2021 Nov 15;45(6):956-970. doi: 10.5993/AJHB.45.6.1. PMID 34969408
- [Background] Whitaker KM, Jones MA, Wallace MK, Catov J, Barone Gibbs B. Associations of objectively measured physical activity and sedentary time with pregnancy-specific health-related quality of life. Midwifery. 2022 Jan;104:103202. doi: 10.1016/j.midw.2021.103202. Epub 2021 Nov 11. PMID 34801955
- [Background] Paley JL, Jones MA, Catov JM, Whitaker KM, Kozai AC, Barone Gibbs B. Associations of Physical Activity and Sedentary Behaviors with Depressive Symptoms and Mood Disturbance Throughout Pregnancy. J Womens Health (Larchmt). 2024 Aug;33(8):1128-1138. doi: 10.1089/jwh.2023.0419. Epub 2024 Feb 6. PMID 38324012
- [Background] Jones MA, Whitaker KM, Paley JL, Thrower A, Stoner L, Barone Gibbs B. Brachial-femoral pulse wave velocity in 2-4-year-old children: a feasibility study. Blood Press Monit. 2023 Feb 1;28(1):11-16. doi: 10.1097/MBP.0000000000000622. Epub 2022 Nov 1. PMID 36606476
- [Background] Jones MA, Whitaker KM, Taverno Ross SE, Davis K, Libertus K, Barone Gibbs B. Maternal Sedentary Behavior and Physical Activity across Pregnancy and Early Childhood Motor Development. Children (Basel). 2021 Jun 25;8(7):549. doi: 10.3390/children8070549. PMID 34201936
- [Background] Jones MA, Whitaker K, Taverno Ross SE, Davis K, Libertus K, Gibbs BB. Maternal Sedentary Behavior and Physical Activity across Pregnancy and Early Childhood Growth. Child Obes. 2022 Sep;18(6):399-408. doi: 10.1089/chi.2021.0202. Epub 2022 Feb 2. PMID 35108109
- [Background] Jones MA, Diesel SJ, Gibbs BB, Whitaker KM. Concurrent Agreement Between ActiGraph and activPAL for Measuring Physical Activity in Pregnant Women and Office Workers. J Meas Phys Behav. 2022 Jun;5(2):69-75. doi: 10.1123/jmpb.2021-0050. Epub 2022 Apr 23. PMID 36340243
- [Background] Whitaker KM, Jones MA, Smith K, Catov J, Feghali M, Kline CE, Santillan M, Santillan D, Zimmerman B, Gibbs BB. Study Design and Protocol of the Multisite Pregnancy 24/7 Cohort Study. Am J Epidemiol. 2024 Feb 5;193(3):415-425. doi: 10.1093/aje/kwad208. PMID 37939072